CLINICAL TRIAL: NCT06207968
Title: Post Market Clinical Follow-up of Knee Surgery Using FH ORTHO SAS Medical Devices (FH ORTHO SAS Knee Observatory)
Brief Title: FH ORTHO SAS Knee Observatory
Status: Not yet recruiting | Type: Observational
Sponsor: FH ORTHO (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-02
Record Dates: First submitted 2023-12-19; First posted 2024-01-17 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Knee Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arthroplasty: Knee prostheses are intended for patients suffering from functionally serious diseases of the knee causing daily disability that is insufficiently improved by medical treatment.
  The functional diseases are among:
  * Knee osteoarthrosis
  * Osteonecrosis of the knee
  * Inflammatory disease
  * Patellofemoral arthritis
  The patients having benefited from an arthroplasty will be followed for at least 15 years (until 20 years).
  Interventions: Device: Knee surgery with FH Ortho devices
- Ligament reconstruction: Ligament reconstruction surgery should be considered for patient who have undergone a rupture of the anterior and/or posterior cruciate ligaments requiring partial or total reconstruction.
  The patients having benefited from a ligament reconstruction will be followed for at least 5 years.
  Interventions: Device: Knee surgery with FH Ortho devices

INTERVENTIONS:
Device: Knee surgery with FH Ortho devices — This clinical investigation is a real-life observatory designed to collect long-term clinical data on patients who have undergone knee joint replacement or knee ligament reconstruction.
  In this type of intervention, one or more medical devices distributed by FH ORTHO SAS may be used by surgeons.

SUMMARY:
The objective of this observatory is to generate additional real life clinical data in accordance with local regulation (i.e. Post-Market Clinical Follow-up (PMCF) study, a study carried out following the European Conformity (CE) marking of a device and intended to answer specific questions relating to clinical safety or performance (i.e. residual risks) of a device when used in accordance with its approved instructions for use (IFU).

The difficulty of such an observatory is to be able to collect data on the different versions of the devices, on the different possible combinations of implants of an knee arthroplasty. The observatory must also be able to cover devices used in ligament reconstruction surgery.

The observatory will be based on the principle of a "dynamic" cohort during the inclusion period, i.e. with possible inclusions to replace the premature exits.

Technical solutions will be implemented to facilitate data collection from surgeons (electronic Case Report Form (eCRF) and from patients (Electronic Patient Reported Outcome (ePRO) on smartphone/tablet/computer) when feasible.

The data to be collected and the different follow-up times are based on our state-of-the-art, clinical evaluation plans and clinical evaluation reports.

DETAILED DESCRIPTION:
PMCF as part of CE mark renewal, to answer questions related to the safety and clinical performance of the devices, when used according to their approved instructions for use.

This is an European, prospective and retrospective, multicenter, non-comparative study.

Randomization is considered impossible due to surgeon preference, anatomical conditions and other patient factors, and the use of different techniques.

This observatory is non-comparative, due to the absence of a gold standard and the technical, logistical and contractual constraints involved.

This PMCF study (CE-marked MD, any class, used as intended) provide additional non-burdensome and non-invasive procedures.

The Observatory will therefore be based on the principle of a "dynamic" cohort, i.e. with possible exits and inclusions throughout the Observatory period.

The aim of this methodology is to have a sufficient number of patients to be able to carry out descriptive statistical analyses each year, and to be able to calculate the evaluation criteria with the longest possible follow-up of results. Data will be collected before surgery, during surgery and at follow-up visits. Data collection will focus on obtaining short- and long-term data for performance and safety evaluation (up to 20 years for knee arthroplasty prostheses; up to 5 years for knee ligament reconstruction devices). In the case of knee arthroplasty, it is recommended to have performance and safety data at 1, 2, 5 and 10 years of follow-up, as well as safety data at 15 and 20 years if possible. In the case of ligament reconstruction, it is recommended to have performance and safety data at 1 and 2 years, as well as safety data at 5 years. The platform will be able to send automatic notifications to surgeons to remind them of scheduled patient follow-ups, missing data, and encourage them to include new patients if necessary. Self-questionnaires will be completed by patients via a web-based platform, available on computer or smartphone/tablet. Alternatively, patients will complete paper self-questionnaires, which will then be entered into the database by the investigating team.

It will also be possible to arrange for direct telephone contact with patients by an independent structure guaranteeing non-dissemination of nominative data (e.g. CRO). Telephone contact can also be made if the patient is geographically remote or has difficulty travelling. Patient recruitment: Continuous, consecutive, prospective and retrospective (for some implants because few implants have been used for this condition) recruitment to guarantee a minimum number of patients per type of device. Individual written information for each patient will be mandatory. A signed patient consent form will be required in Europe, after sufficient time for reflection.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing or having undergone implantation of medical devices distributed by FH ORTHO SAS for knee arthroplasty and ligament reconstruction, used in accordance with their approved IFU, in one of the centers participating in the Observatory.
* Patient is at least 18 years old at the time of surgery
* Patient agreeing to participate after having been informed orally and in writing (with written consent if required locally)
* In some countries, such as France, the patient will have to be socially insured to be included in the study.

Exclusion Criteria:

For Arthroplasty:

1. Infection, or latent infection
2. A mental or neuromuscular disorder that might create an unacceptable risk of instability, prosthetic fixation failure, or complications after surgery
3. Insufficient bone stock for proper implant fixation
4. It is the surgeon's responsibility to make sure that the patient does not have any known allergies to one of the compounds of the material listed on the product label.
5. Metabolic diseases that might compromise bone regrowth
6. Drug addiction
7. Incomplete bone growth

For Ligament reconstruction:

1. Infection, or latent infection
2. A mental or neuromuscular disorder that might create an unacceptable risk of instability, prosthetic fixation failure, or complications after surgery
3. Insufficient bone stock
4. Known allergies to one of the compounds of the material listed on the product label.
5. Metabolic diseases that might compromise bone regrowth
6. Uncooperative patient unable to follow recommendations

As the medical devices are used in real life according to their indications, pregnant or breastfeeding women are not excluded from the study, but for safety reasons it is not advisable to include them in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will be representative of the target population of the medical devices.
  The aim is to recruit in the first 3 years in 15-20 sites in France, 487 patients who have benefited from knee arthroplasty or ligament reconstruction of the knee.
  Arthroplasty arm: Knee prostheses are intended for patients suffering from functionally serious diseases of the knee causing daily disability that is insufficiently improved by medical treatment (Knee osteoarthrosis, Osteonecrosis of the knee, Inflammatory disease, or Patellofemoral arthritis).
  Ligament reconstruction arm: Ligament reconstruction surgery should be considered for patient who have undergone a rupture of the anterior and/or posterior cruciate ligaments requiring partial or total reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 487 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2044-06 (Estimated); Study Completion 2044-06 (Estimated)

PRIMARY OUTCOMES:
Revision rate | 2 months, 3-6 months, 1 year, 2 years, 5 years, 10 years, 15 years, 20 years
  Evaluate the revision rate at the longest follow-up possible for arthroplasty arm
Revision rate | 2 months, 3-6 months, 1 year, 2 years, 5 years
  Evaluate the revision rate at the longest follow-up possible for ligament reconstruction arm

SECONDARY OUTCOMES:
International Knee Society (IKS 2011) score | Pre-operative, 3-6months, 1 year, 2 years, 5 years, 10 years
  Mobility, Pain and Function for Arthroplasty arm.
  It includes a 100-point objective score and a subjective score made up of 3 domains evaluating satisfaction on 40 points, patient expectations on 15 points using different items between the pre- and post-operative phases, as well as functional activities on 100 points. The total score was 255 points. There are no levels and the results are expressed as raw scores. Higher scores mean a better outcome.
Complications/Adverse events | During surgery, Immediate (0-2months), 3-6months, 1 year, 2 years, 5 years, 10 years
  any adverse events leading or not to re-intervention (with or without change of the implant), including device malfunctions
International Knee Documentation Committee (IKDC 2000) score | Pre-operative, 1 year, 2 years
  Mobility, Pain and Function for Ligament Reconstruction arm
  This self-questionnaire is divided into three parts (symptoms, sporting activities, function) and gives a score between 0 (worst) and 100 (best). This score is interpreted as a measure of functional capacity, with the highest scores representing the best levels of function and the lowest levels representing symptoms. A score of 100 means that there are no limits to daily activities and sports and that symptoms are non-existent.
Lysholm Knee Scoring Scale | Pre-operative, 1 year, 2 years
  Mobility, Pain and Function for Ligament Reconstruction arm The Lysholm Knee Score is a questionnaire that the patient completes with the therapist. The questionnaire is designed to assess the degree of knee instability, in terms of both impairment and limitation.
  The Lysholm Knee Score calculates and rates an overall score from 0 to 100 based on 8 domains: squatting, locking, pain, stair climbing, weight bearing, instability and oedema. Doctors use this condition-specific subjective outcome score to assess a patient's progress after knee surgery or injury. Scores between 95 and 100 are considered exceptional, those between 84 and 94 acceptable, those between 65 and 83 fair and those below 65 poor.
Tegner activity level scale | Pre-operative, 1 year, 2 years
  Mobility, Pain and Function for Ligament Reconstruction arm
  The Tegner activity scale is a numerical scale with values ranging from 0 to 10, each representing a different activity. A person is considered to have an activity level of 10 if they play highly competitive sports such as rugby, football and soccer. A person who plays the above sports recreationally is considered to have an activity level of 6. A person with knee problems who is on sick leave or receiving a disability pension is considered to have an activity level of 0.
Knee laxity (clinical section) | Pre-operative, 3-6 months
  Mobility, Pain and Function for Ligament Reconstruction arm.
  This questionnaire is completed by the physician. He will assessed laxity of operated knee, as:
  Pivot Shift test: absent (0), grade 1 (+), grade 2 (++), grade 3 (+++).
Complications/Adverse events | During surgery, Immediate (0-2months), 3-6months, 1 year, 2 years, 5 years
  Any adverse events leading or not to re-intervention (with or without change of the implant), including device malfunctions
Visual Analogue Scale (VAS) | 1 year, 2 years, 5 years, 10 years, 15 years, 20 years
  for arthroplasty arm Pain rating scale. A straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the pain to be measured orientated from the left (worst) to the right (best).
  The scale is given to the patient during the consultation, the patient indicates his/her level of pain and the surgeon then transcribes the score.
Visual Analogue Scale (VAS) | 1 year, 2 years, 5 years
  for ligament reconstruction arm Pain rating scale. A straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the pain to be measured orientated from the left (worst) to the right (best).
  The scale is given to the patient during the consultation, the patient indicates his/her level of pain and the surgeon then transcribes the score.
ASA (American Society of Anesthesiologists)-score | Pre-operative
  The American Society of Anesthesiologists proposes five classes of patients requiring anaesthesia.
  Class 1: patient in good health. Class 2: patient with moderate general illness. Class 3: patient with a serious but not incapacitating general illness. Class 4: patient with a life-threatening general illness. Class 5: a moribund patient who would not survive 24 hours without the procedure, the outcome of which is uncertain.

OTHER OUTCOMES:
Patient satisfaction | 3-6months, 1 year, 2 years, 5 years, 10 years
  A simple questionnaire consisting of 3 questions will be proposed to the patient. The 2 first one will be to graduate the satisfaction regarding the mobility and the pain of the operated knee and the last one is the yes/No question regarding the surgery reiteration.
X-ray | 3-6months
  check the position of the prosthesis using medical imaging. Desired position: Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Charles KAJETANEK, MD, Principal Investigator — Hôpitaux Privés Rennais - Saint-Grégoire (Vivalto Santé) Institut Locomoteur de l'Ouest
Locations (10):
- France (10):
  - Clinique De La Chataigneraie, Beaumont
  - Clinique De La Miotte, Belfort
  - Polyclinique St Privat, Boujan-sur-Libron
  - Clinique Du Val D'Ouest, Écully
  - C.H. Raymond Poincare, Garches
  - Hôpital Saint Vincent de Paul, Lille
  - Hôpital Prive St Grégoire, Saint-Grégoire
  - Polyclinique De L'Europe, Saint-Nazaire
  - Medipole Garonne, Toulouse
  - Hôpital Privé Océane, Vannes

IPD SHARING:
Plan to Share IPD: No